CLINICAL TRIAL: NCT04719130
Title: Effectiveness of Multimodal Circuit Exercises for Chronic Musculoskeletal Pain in Older Adults: a Randomized Controlled Trial Protocol
Brief Title: Multimodal Circuit Exercises for Chronic Musculoskeletal Pain in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Federal University of Minas Gerais (Other); Federal University of Tocantins (Unknown); Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNB11121
Record Dates: First submitted 2021-01-12; First posted 2021-01-22 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2021-01

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: Exercise Therapy; Multimodal exercise
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel study (two arms) with blinded outcome assessments.
Who Masked: Outcomes Assessor
Masking Description: Another researcher collaborator (blinded) will be carried out the outcomes investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Will received multimodal circuit exercise group.
  Interventions: Other: Multimodal circuit exercise
- Control Group (Active Comparator): Will received multidisciplinary lectures on pain and usual care provided by the Basic Health Units.
  Interventions: Other: Multidisciplinary lectures

INTERVENTIONS:
Other: Multimodal circuit exercise — A structured and supervised multimodal exercise circuit twice a week, under 12 weeks program. The circuit workout program consists of 8 exercises, divided into motor coordination, balance, strength, and aerobic exercises. The exercises will be employed in a reserved room inside of the Basic Health Units. The sessions of exercises will last approximately 50 minutes,
  Arms: Experimental Group
Other: Multidisciplinary lectures — Multidisciplinary lectures on pain and usual care provided by the Basic Health Units. A cycle of multidisciplinary lectures on pain will be offered by professionals in physical education, nursing, physiotherapy, medicine, psychology and social work that will take place in the Basic Health Units every 15 days.
  Arms: Control Group

SUMMARY:
Analyze the effectiveness of a multimodal circuit exercise program on chronic musculoskeletal pain and disability in older adults.

DETAILED DESCRIPTION:
This is a randomized parallel study (two arms) with blinded outcome assessments. The participants' recruitment will be done by a non-probabilistic sampling resulting from invitations to Basic Health Units. The sample size estimation indicated 164 participants. Participants will be allocated, by means of a randomization process, to one of two groups (82 for each group): Experimental Group (multimodal circuit exercise) or Control Group (cycle of multidisciplinary lectures on pain ). The primary outcomes are global chronic pain intensity and global functional disability scores. The secondary outcomes are functional mobility and cardiorespiratory capacity. All analyses will be processed using the RStudio software. The differences will be considered statistically significant when a 2-tailed p-value is less than 5% (p < 0.05). The statistical analysis will follow the intention to treat. Discussion: This study will discuss the effects of multimodal circuit exercise on global chronic pain intensity and global body functional disability scores. The hypothesize is that multimodal exercises will reduce musculoskeletal chronic pain and disability in older adults to the same extent as traditional supervised and structured exercises.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from both sexes;
* Aged 60 or higher;
* Had a history of chronic pain in at least one synovial joint for more than three months.

Exclusion Criteria:

* Participants with some types of co-morbidities that may interfere with the research parameters, such as a history of stroke, stenosis of the spinal canal, severe heart disease, fibromyalgia, rheumatoid arthritis;
* Participants who presented a level of pain between 7 and 10 points on the Numeric Rate Scale (NRS) in any body location;
* Participants being under psychiatric treatment with sensory deficits (visual, auditory and intellectual)
* Participants performing any supervised and structured exercise at the moment of study enrollment or six months before.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Change on pain intensity. | Change from Baseline at immediately post-intervention
  Will be used the Brief Pain Inventory (BPI). The Brief Pain Inventory (BPI) [32, 33]- a multidimensional, easily used questionnaire, aiming to diagnose a patient's chronic pain during the last 24 hours, categorized into 11 questions, scaled from 0 to 10, in which 10 indicates "worst pain imaginable".
Change on disability. | Change from Baseline at immediately post-intervention
  Will be used the Independence Index in Activities of Daily Living (Katz Index - KI). The total KI score is in the range 0 to 6, whose score 6 represents an independent patient and 0 indicates a highly dependent patient.
Change on pain intensity. | Change from Baseline at immediately post-intervention
  Will be used the Numeric Rating Scale. It is a subjective procedure, widely used due to its reliability, as the patients classify their pain at the moment within a scale from 0 (no pain at all) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Change on cardiorespiratory capacity. | Change from Baseline at immediately post-intervention
  Will be used the 6-minute walk test.
Change on functional mobility | Change from Baseline at immediately post-intervention
  Will be used the Time up and go test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The excel data-base will be shared with all data when the manuscript were submitted to a peer-review process. If published, the paper will be provided all data base by supplementary material.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The excel data-base will be shared with all data when the manuscript were submitted to a peer-review process. If published, the paper will be provided all data base by supplementary material.

REFERENCES:
- [Background] Blyth FM, Noguchi N. Chronic musculoskeletal pain and its impact on older people. Best Pract Res Clin Rheumatol. 2017 Apr;31(2):160-168. doi: 10.1016/j.berh.2017.10.004. Epub 2017 Nov 4. PMID 29224694
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. 2015 Feb 18;350:h444. doi: 10.1136/bmj.h444. PMID 25694111
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Derived] Ribeiro DBG, Gentil PRV, Resende RA, Carregaro RL, Fonseca STD, Martins WR. Effectiveness of multimodal circuit exercises for chronic musculoskeletal pain in older adults: A randomized controlled trial protocol. J Frailty Sarcopenia Falls. 2022 Sep 1;7(3):175-182. doi: 10.22540/JFSF-07-175. eCollection 2022 Sep. PMID 36119552